CLINICAL TRIAL: NCT00036101
Title: Study of Aripiprazole in the Treatment of Patients With Acute Symptoms in Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Purpose: Treatment
Other Study IDs: CN138-074
Record Dates: First submitted 2002-05-07; First posted 2002-05-09 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2007-09

CONDITIONS: Bipolar Disorder
Keywords: Bipolar I Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Aripiprazole

INTERVENTIONS:
Drug: aripiprazole

SUMMARY:
The purpose of this study is to learn if aripiprazole is effective for the treatment of patients with acute symptoms of Bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

Patients with acute symptoms of Bipolar Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-02; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Local Institution, Tuscaloosa, Alabama
  - Local Institution, Little Rock, Arizona
  - Local Institution, Beachwood, California
  - Local Institution, Chula Vista, California
  - Local Institution, Riverside, California
  - Local Institution, San Clemente, California
  - Local Institution, San Diego, California
  - Local Institution, Stanford, California
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, North Miami, Florida
  - Local Institution, Winter Park, Florida
  - Local Institution, Honolulu, Hawaii
  - Local Institution, Chicago, Illinois
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Louisville, Kentucky
  - Local Institution, Belmont, Massachusetts
  - Local Institution, Newton Center, Massachusetts
  - Local Institution, New Baltimore, Michigan
  - Local Institution, Lawrence, New York
  - Local Institution, Butner, North Carolina
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Medina, Ohio
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Austin, Texas
  - Local Institution, Houston, Texas
  - Local Institution, Falls Church, Virginia
  - Local Institution, Bellevue, Washington